CLINICAL TRIAL: NCT07255651
Title: Effect of Transfer Energy Capacitive and Resistive Therapy on Pain and Range of Motion After Flexor Tendon Repair
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Basma Rajai Amer Amer, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P.T.REC/012/006005
Record Dates: First submitted 2025-11-20; First posted 2025-12-01 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Flexor Tendon Rupture
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transfer Energy Capacitive and Resistive (TECAR) therapy + Early mobilization protocol (Experimental): It will receive Transfer Energy Capacitive and Resistive (TECAR) therapy in addition to early mobilization protocol for a month.
  Interventions: Device: Transfer Energy Capacitive and Resistive (TECAR) therapy; Other: Early mobilization protocol
- Early mobilization protocol (Active Comparator): It will receive their early mobilization protocol only for a month.
  Interventions: Other: Early mobilization protocol

INTERVENTIONS:
Device: Transfer Energy Capacitive and Resistive (TECAR) therapy — Before each session, cables will be checked, the therapist will explain the procedure, the patient will be positioned comfortably, and conductive cream will be applied. The active electrode will be moved in circular motions over the injured tendon while the inactive electrode will be placed under the forearm. Intensity will be set to a comfortable, moderate level based on patient sensation. Radio-frequency (RF) energy will be delivered via capacitive mode for 2 minutes per digit, then resistive mode for 4 minutes per digit (total 6 minutes per digit). Treatment will include 8 sessions, twice weekly.
  Arms: Transfer Energy Capacitive and Resistive (TECAR) therapy + Early mobilization protocol
Other: Early mobilization protocol — The dorsal splint/cast will position the wrist at neutral or 15-30° extension with metacarpophalangeal (MCP) joints at 70-90° flexion, featuring low edges for exercise without removal. It will be worn full-time for the first 3 weeks post-surgery, then based on environmental safety (only during sleep and outside home if safe) for weeks 4-6. Patients will begin outpatient physical therapy from week 1 with active mobilization and home exercises every 2 hours. Dressings will be changed every other day. During weeks 1-2, passive/active flexion/extension will follow the Duran protocol (25-50% range of motion) with splint worn during therapy. Weeks 3-4 will progress to 75-100% range of motion, with splint removal at week 4 for active tenodesis exercises. Weeks 5-6 will add tendon gliding, blocking exercises, and light activities while avoiding strenuous lifting or gripping. This progressive protocol will ensure safe healing while gradually restoring function.

SUMMARY:
The purpose of this study is to evaluate the impact of Transfer Energy Capacitive and Resistive therapy (TECAR) on pain and range of motion (ROM) after hand flexor tendon repair.

DETAILED DESCRIPTION:
Lacking satisfactory healing of intrasynovial tendons, such as the flexor tendons of the hand, is particularly challenging due to the formation of fibrous adhesions between the tendon, sheath and surrounding tissues which can further limit mobility.

Transfer Energy Capacitive and Resistive therapy (TECAR) enhances the body's natural ability to repair tissues and reduce pain by improving blood flow and promoting additional benefits, such as cell proliferation. This process, primarily linked to the flow of current, supports cell growth and plays a significant role in the healing process.

There is a lack in quantitative knowledge and information in the published studies about the benefits of TEcar therapy on the improvement of hand function after long flexor tendon repair . So, this study is designed to outline the therapeutic impact of TEcar therapy on pain and ROM after hand flexor tendon repair.

ELIGIBILITY:
Inclusion Criteria:

* Ages of patients will be ranged from 20 to 35 years.
* All patients underwent flexor tendon primary direct repair
* All patients will be referred by a surgeon before starting the study procedure.

Exclusion Criteria:

* Patient with digital nerve repairs.
* Patients with associated vascular injuries requiring arterial repair.
* Patients with associated crush injuries and soft tissue loss.
* Patients with associated bone fractures.
* Patients with associated extensor tendon injuries .
* Patients with preexisting problems limiting joint motion.
* Patients with diminished cognitive capacity.
* Patients with history of previously failed repair.
* Patients with allergic reactions to certain substances in the conductive cream
* Patients with sensation impairment .

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-15 (Estimated)

PRIMARY OUTCOMES:
Active range of motion (ROM) of the proximal interphalangeal (PIP) joint | one month
  Active ROM of the PIP joint will be assessed, at the 2nd, 4th, and 6th postoperative weeks using a finger goniometer, with the patient sitting, forearm mid-position and supported on a plinth. The therapist will stabilize the metacarpophalangeal (MCP) joint in 90° flexion at the injured phalanx. The goniometer's axis will be placed over the upper surface of the PIP joint, with the stationary arm aligned to the proximal phalanx's longitudinal axis and the movable arm aligned to the middle phalanx's longitudinal axis. The patient will be instructed to actively flex and then extend the PIP joint through its full range (normally 0°-100°), and the measured ROM will be recorded.
Active range of motion (ROM) of the distal interphalangeal (DIP) joint | one month
  Active ROM of the DIP joint will be assessed with the patient seated, forearm in mid-position and supported on the plinth. From a neutral wrist position, the therapist will stabilize the metacarpophalangeal (MCP) joint in 90° flexion and the middle phalanx in extension. The goniometer axis will be placed over the upper surface of the DIP joint, with the stationary arm aligned to the middle phalanx's longitudinal axis and the movable arm aligned to the distal phalanx. The patient will actively flex and extend the DIP joint through its full range (0°-90°), and the ROM will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Hsham Mahran, PhD, Study Chair — Professor, Cairo university; Ahmed Mahmoud Ali Gabr Zarraa, PhD, Study Director — Lecturer, Cairo university; Amr Abdallah Gomaa, PhD, Study Director — Assistant Professor, Suez Canal university
Locations (1):
- Suez Canal University Hospital, Ismailia, Egypt